CLINICAL TRIAL: NCT04588935
Title: To Develop and Implement a Method for Medical Prevention of Cardiovascular Diseases Caused by Complex Treatment of Patients With Primary Operated Breast Cancer
Brief Title: Prevention of Cardiovascular Diseases Caused by Complex Treatment of Patients With Primary Operated Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State Institution "Republican Scientific and Practical Center" Cardiology, Belarus (Other)
Responsible Party: Principal Investigator, Dr. Chernyak Sergey, Researcher, Hypertension Laboratory Republican Scientific and Clinical Cardiology Center Republic of Belarus, Belarus, State Institution "Republican Scientific and Practical Center" Cardiology, Belarus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20192755
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Women With Breast Cancer
MeSH Terms: interventions — Bisoprolol; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): women with breast cancer, with a morphologically confirmed diagnosis before the appointment of anticancer therapy, untreated
- Group 2 (Active Comparator): women with breast cancer, with a morphologically confirmed diagnosis before the appointment of anticancer therapy, receiving treatment with a combination of bisoprolol and perindopril
  Interventions: Drug: Bisoprolol; Perindopril;

INTERVENTIONS:
Drug: Bisoprolol; Perindopril; — based on the results of the patient study, different drug therapy regimens for cardiovascular complications during chemotherapy will be proposed
  Other Names: Bisoprolol; Perindopril
  Arms: Group 2

SUMMARY:
To develop a method of medical prevention of cardiovascular diseases caused by cardiotoxicity against the background of complex treatment of patients with primary resectable breast cancer to reduce the risk of cardiovascular complications

DETAILED DESCRIPTION:
Purpose of the study: to develop a method of medical prevention of cardiovascular diseases caused by cardiotoxicity against the background of complex treatment of patients with primary resectable breast cancer to reduce the risk of cardiovascular complications

ELIGIBILITY:
Inclusion Criteria:

* women with breast cancer, with a morphologically confirmed diagnosis before the appointment of anticancer therapy.

Exclusion Criteria:

* presence of other oncological diseases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
development of cardiovascular diseases and complications | 4 years
  hypertension, cardiomyopathy, arrhythmia's, myocardial infarction, heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific and Practice Center of Cardiology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No